CLINICAL TRIAL: NCT05819879
Title: Peri Capsular Nerve Group Block Versus Sciatico Femoral Block to Assess the Incidence of Post Amputation Syndroms in Patients Undergoing Above Knee Amputation Surgeries
Brief Title: PENG Block vs Sciatico Femoral Block in the Incidence of Post Amputation Syndroms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ahmed Ibrahim Hussien Hussien, Resident of Anesthesia, Surgical Intensive Care and Pain Medicine, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AP2102-30101
Record Dates: First submitted 2023-03-07; First posted 2023-04-19 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Femoral Nerve Block; Amputation of Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG group (Active Comparator)
  Interventions: Procedure: peri capsular nerve group block
- scaitico femoral block group (Active Comparator)
  Interventions: Procedure: scaitico femoral block

INTERVENTIONS:
Procedure: peri capsular nerve group block — The block will be administered under ultrasound guidance with low frequency curvilinear probe. The probe will be placed parallel to the inguinal crease, at the level of anterior superior iliac spine. The scanning will be done with gradual caudad movement of the probe. After the anterior inferior iliac spine (AIIS) become visible, the probe will be turned slightly medial until the hyperechoic continuous shadow of superior pubic ramus become visible. The psoas muscle with prominent tendon will be identified just above the pubic ramus. The target is the plane between these two structures. Aligning the pubic ramus in the center of the image and targeting the pubic ramus just medial to the AIIS, a standard 25G Quincke needle will be introduced and 20 mL 0.125% bupivacaine with 4 mg dexamethasone was administered using ultrasound-guided out-of-plane technique.
  Arms: PENG group
Procedure: scaitico femoral block — . After draping the left inguinal region, the femoral nerve will be identified lateral to the femoral artery using a 5- to 13-MHz linear phased array transducer ). Under ultrasound guidance, a 25G Quincke needle will be introduced toward the femoral nerve parallel to the ultrasound beam, and 20 mL of a local anesthetic mixture 20 mL 0.125% bupivacaine with 4 mg dexamethasone will be injected. The trajectory of the needle was adjusted to achieve even distribution of the local anesthetics around the femoral nerve. Then, the patient will be placed in the right lateral position with the left hip and knee joints flexed by 30° to 50°. Following the identification of the left sciatic nerve located in the intermuscular plane of the gluteus maximus and medius muscles between the ipsilateral ischial tuberosity and greater trochanter using a convex phased array transducer 20 mL 0.125% bupivacaine with 4 mg dexamethasone will be placed near the sciatic nerve through the 22-ga Tuohy needle
  Arms: scaitico femoral block group

SUMMARY:
assess the effectiveness of peri-capsular nerve group block and scaitico femoral block in the incidence of post amputation syndrome in patients undergoing above knee amputation.

DETAILED DESCRIPTION:
The loss of a body part can lead to pain and other sensations that fall into three distinct descriptive categories, namely phantom sensations, phantom pain, and residual pain. Phantom sensations are defined as pain-free perceptions emanating from the lost body part after deafferentation, and phantom pain is a painful or unpleasant sensation in the distribution of the lost or deafferented body part 5. Phantom sensations can be a different expression of phantom pain and interfere with rehabilitation therapy by enhancing and interacting with phantom pain.

The current standard of care is pre-operative nerve blockade to prevent peripheral sensitization leading to future onset of phantom limb pain. Successful outcomes necessitate effective communication between the surgeon, anesthesiologist, and the various teams involved in the post-operative rehabilitation of the patient. A consultation with the Acute Pain Service or similar entity that performs peripheral nerve blockade pre-operatively and then follows the patient during their post-operative inpatient course is an important factor in the success in early prevention of acute and chronic pain for these patients.

Pericapsular nerve group block or PENG block is a novel regional nerve block to provide analgesia in fractured hip patients. It is primarily an ultrasound-guided (USG) technique where target area is the pelvic rim (superior pubic ramus) near iliopectineal eminence, deep to fascia of iliopsoas muscle. Articular branches of femoral nerve and accessory obturator nerves, which cross over the bony rim, are primary targets of the PENG block.however, by increasing volume of local anesthetic drug; other nerves (obturator, femoral, genitofemoral, and lateral femoral cutaneous nerve) can be blocked.

This block is a new regional anesthesia technique based on blocking the femoral nerve (FN) and accessory obturator nerve (ON) with a single injection.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I and II
* Age above 20 and less than 60 years.
* Patients undergoing above knee amputation due to any type of cancer

Exclusion Criteria:

* Patient refusal.
* Local infection at the puncture site.
* Coagulopathy.
* Cognitive disorders.
* Unstable cardiovascular disease.
* History of psychiatric disorders.
* History of drug abuse.
* Patients allergic to medication used.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of the efficacy of peri capsular nerve group block | 24 hours postoperatively
  Incidence of the efficacy of peri capsular nerve group block in reducing the post amputation limb pain for 24h and to compare it with the efficacy of scaitico femoral nerve block in reducing the post amputation limb pain as well.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Ibrahim Hussien Hussien, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the principal investigator
Supporting Information: Study Protocol
Time Frame: One year